CLINICAL TRIAL: NCT06039371
Title: SPECTRA: Supraphysiological Androgen to Enhance Treatment Activity
Brief Title: Supraphysiological Androgen to Enhance Treatment Activity in Metastatic Castration-Resistant Prostate Cancer, SPECTRA Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RG1123642; NCI-2023-05597 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); FHIRB0020106 (Other: Fred Hutch/University of Washington Cancer Consortium); 2P50CA097186 (NIH)
Record Dates: First submitted 2023-08-21; First posted 2023-09-15 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Castration-Resistant Prostate Carcinoma; Metastatic Prostate Adenocarcinoma; Stage IVB Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Biopsy; Specimen Handling; Carboplatin; Etoposide; testosterone 17 beta-cypionate; Testosterone Propionate; Methyltestosterone; Absorptiometry, Photon; Magnetic Resonance Spectroscopy; X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Cohort Ia (testosterone cypionate, carboplatin) (Active Comparator): Patients continue to receive ADT per standard of care and receive testosterone cypionate IM on day 1 of cycle 1. Patients then receive testosterone cypionate IM and carboplatin IV on day 1 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. All patients undergo a biopsy, blood sample collection, bone scan and CT scan throughout the study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Bone Scan; Drug: Carboplatin; Procedure: Computed Tomography; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Testosterone Cypionate; Procedure: Dual X-ray Absorptiometry
- Cohort Ib (testosterone cypionate, carboplatin) (Active Comparator): Patients continue to receive ADT per standard of care and receive carboplatin IV on day 1 of cycle 1. Patients then receive testosterone cypionate IM and carboplatin IV on day 1 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. All patients undergo a biopsy, blood sample collection, bone scan and CT scan throughout the study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Bone Scan; Drug: Carboplatin; Procedure: Computed Tomography; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Testosterone Cypionate; Procedure: Dual X-ray Absorptiometry
- Cohort Ic (testosterone cypionate, carboplatin) (Experimental): Patients continue to receive ADT per standard of care and receive testosterone cypionate IM and carboplatin IV on day 1 of cycle 1. Patients then receive testosterone cypionate IM and carboplatin IV on day 1 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. All patients undergo a biopsy, blood sample collection, bone scan and CT scan throughout the study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Bone Scan; Drug: Carboplatin; Procedure: Computed Tomography; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Testosterone Cypionate; Procedure: Dual X-ray Absorptiometry
- Cohort IIa (testosterone cypionate, etoposide) (Active Comparator): Patients continue to receive ADT per standard of care and receive testosterone cypionate IM on day 1 of cycle 1. Patients then receive testosterone cypionate IM on day 1 and etoposide PO QD on days 1-14 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. All patients undergo a biopsy, blood sample collection, bone scan and CT scan throughout the study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Drug: Etoposide; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Testosterone Cypionate; Procedure: Dual X-ray Absorptiometry
- Cohort IIb (testosterone cypionate, etoposide) (Active Comparator): Patients continue to receive ADT per standard of care and receive etoposide PO QD on days 1-14 of cycle 1. Patients then receive testosterone cypionate IM on day 1 and etoposide PO QD on days 1-14 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. All patients undergo a biopsy, blood sample collection, bone scan and CT scan throughout the study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Drug: Etoposide; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Testosterone Cypionate; Procedure: Dual X-ray Absorptiometry
- Cohort IIc (testosterone cypionate, etoposide) (Experimental): Patients continue to receive ADT per standard of care and receive testosterone cypionate IM on day 1 and etoposide PO QD on days 1-14 of cycle 1. Patients then receive testosterone cypionate IM on day 1 and etoposide PO QD on days 1-14 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. All patients undergo a biopsy, blood sample collection, bone scan and CT scan throughout the study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Drug: Etoposide; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Testosterone Cypionate; Procedure: Dual X-ray Absorptiometry
- Cohort IIIa (ADT, testosterone cypionate, LuPSMA) (Experimental): Patients continue to receive ADT per standard of care and receive testosterone cypionate IM on day 1 of cycles 1-6. Patients receive LuPSMA IV on day 1 of cycles 2-6. Cycles repeat every 6 weeks for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive testosterone cypionate IM on day 1 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. All patients undergo a biopsy on study and blood sample collection on study, and bone scans, DEXA and CT scans throughout the trial. Patients may also undergo an optional second biopsy at the end of study treatment. Patients also undergo 68Ga-PSMA PET at screening and SPECT/CT throughout the study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Testosterone Cypionate; Other: Radioconjugate; Procedure: Dual X-ray Absorptiometry; Other: Gallium Ga 68-PSMA-617; Procedure: Positron Emission Tomography; Procedure: Single Photon Emission Computed Tomography
- Cohort IIIb (ADT, testosterone cypionate, LuPSMA) (Experimental): Patients continue to receive ADT per standard of care and LuPSMA IV on day 1 of cycles 1-6. Patients also receive testosterone cypionate IM on day 1 of cycles 2-6 . Cycles repeat every 6 weeks for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients receive testosterone cypionate IM on day 1 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo 68Ga-PSMA PET at screening and SPECT/CT throughout the study. All patients undergo a biopsy on study and blood sample collection on study, and bone scans, DEXA and CT scans throughout the trial. Patients may also undergo an optional second biopsy at the end of study treatment.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Testosterone Cypionate; Other: Radioconjugate; Procedure: Dual X-ray Absorptiometry; Other: Gallium Ga 68-PSMA-617; Procedure: Positron Emission Tomography; Procedure: Single Photon Emission Computed Tomography
- Cohort IIIc (ADT, testosterone cypionate, LuPSMA) (Experimental): Patients continue to receive ADT per standard of care and receive testosterone cypionate IM on day 1 and LuPSMA IV on day 1 of cycles 1-6. Cycles repeat every 6 weeks for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive testosterone cypionate IM on day 1 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo 68Ga-PSMA PET at screening and SPECT/CT throughout the study. All patients undergo a biopsy on study and blood sample collection on study, and bone scans, DEXA and CT scans throughout the trial. Patients may also undergo an optional second biopsy at the end of study treatment.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Testosterone Cypionate; Other: Radioconjugate; Procedure: Dual X-ray Absorptiometry; Other: Gallium Ga 68-PSMA-617; Procedure: Positron Emission Tomography; Procedure: Single Photon Emission Computed Tomography

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo a biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Scan — Undergo bone scan
  Other Names: Bone Scintigraphy
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
  Arms: Cohort Ia (testosterone cypionate, carboplatin); Cohort Ib (testosterone cypionate, carboplatin); Cohort Ic (testosterone cypionate, carboplatin)
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Drug: Etoposide — Given PO
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP-16; VP-16-213; VP16
  Arms: Cohort IIa (testosterone cypionate, etoposide); Cohort IIb (testosterone cypionate, etoposide); Cohort IIc (testosterone cypionate, etoposide)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Drug: Testosterone Cypionate — Given IM
  Other Names: depAndro; Depo-Testosterone; Depotest; Depovirin; Pertestis; Virilon
Other: Radioconjugate — Given LuPSMA IV
  Other Names: Radio Conjugates
  Arms: Cohort IIIa (ADT, testosterone cypionate, LuPSMA); Cohort IIIb (ADT, testosterone cypionate, LuPSMA); Cohort IIIc (ADT, testosterone cypionate, LuPSMA)
Procedure: Dual X-ray Absorptiometry — Undergo DEXA
  Other Names: BMD scan; bone mineral density scan; DEXA; DEXA scan; dual energy x-ray absorptiometric scan
Other: Gallium Ga 68-PSMA-617 — Given gallium 68Ga-PSMA-617
  Other Names: 2247839-19-4; 68Ga-PSMA-617; Gallium-68 PSMA-617; VIPIVOTIDE TETRAXETAN GALLIUM GA-68
  Arms: Cohort IIIa (ADT, testosterone cypionate, LuPSMA); Cohort IIIb (ADT, testosterone cypionate, LuPSMA); Cohort IIIc (ADT, testosterone cypionate, LuPSMA)
Procedure: Positron Emission Tomography — Undergo 68Ga-PSMA PET
  Other Names: Medical Imaging; PET; PET scan
  Arms: Cohort IIIa (ADT, testosterone cypionate, LuPSMA); Cohort IIIb (ADT, testosterone cypionate, LuPSMA); Cohort IIIc (ADT, testosterone cypionate, LuPSMA)
Procedure: Single Photon Emission Computed Tomography — Undergo SPECT/CT
  Other Names: Medical Imaging; SPECT
  Arms: Cohort IIIa (ADT, testosterone cypionate, LuPSMA); Cohort IIIb (ADT, testosterone cypionate, LuPSMA); Cohort IIIc (ADT, testosterone cypionate, LuPSMA)

SUMMARY:
This phase II trial studies how well giving testosterone at levels higher than normally found in the body (supraphysiological) works to enhance chemotherapy treatment, and Lutetium 177Lu-prostate specific-membrane antigen (PSMA)-617 (LuPSMA) in patients with prostate cancer that has progressed despite being previously treated with androgen therapies and has spread from where it first started (prostate) to other places in the body (metastatic castration-resistant prostate cancer). In patients that have developed progressive cancer in spite of standard hormonal treatment, administering supraphysiological testosterone may result in regression of tumors by causing deoxyribonucleic acid (DNA) damage in tumor cells that have adapted to low testosterone conditions. Carboplatin is in a class of medications known as platinum-containing compounds. Carboplatin works by killing, stopping or slowing the growth of tumor cells. Etoposide is in a class of medications known as podophyllotoxin derivatives. It blocks a certain enzyme needed for cell division and DNA repair and may kill tumor cells. Radioactive drugs, such as LuPSMA, may carry radiation directly to tumor cells and not harm normal cells. Giving supraphysiological levels of testosterone and carboplatin or etoposide or LuPSMA together may be an effective treatment for metastatic castration-resistant prostate cancer.

DETAILED DESCRIPTION:
OUTLINE:

Patients are assigned based on personal preference to 1 of 3 cohorts.

COHORT I: Patients are then assigned to 1 of 3 sub-cohorts within cohort I.

COHORT Ia: Patients continue to receive ADT and receive testosterone cypionate intramuscularly (IM) on day 1 of cycle 1. Patients then receive testosterone cypionate IM and carboplatin intravenously (IV) on day 1 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

COHORT Ib: Patients continue to receive ADT and receive carboplatin IV on day 1 of cycle 1. Patients then receive testosterone cypionate IM and carboplatin IV on day 1 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

COHORT Ic: Patients continue to receive ADT and receive testosterone cypionate IM and carboplatin IV on day 1 of cycle 1. Patients then receive testosterone cypionate IM and carboplatin IV on day 1 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

COHORT II: Patients are then assigned to 1 of 3 sub-cohorts within cohort II.

COHORT IIa: Patients continue to receive ADT and receive testosterone cypionate IM on day 1 of cycle 1. Patients then receive testosterone cypionate IM on day 1 and etoposide orally (PO) once daily (QD) on days 1-14 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

COHORT IIb: Patients continue to receive ADT and receive etoposide PO QD on days 1-14 of cycle 1. Patients then receive testosterone cypionate IM on day 1 and etoposide PO QD on days 1-14 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

COHORT IIc: Patients continue to receive ADT and receive testosterone cypionate IM on day 1 and etoposide PO QD on days 1-14 of cycle 1. Patients then receive testosterone cypionate IM on day 1 and etoposide PO QD on days 1-14 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

COHORT III: Patients are assigned to 1 of 3 sub-cohorts within cohort III.

COHORT IIIa: Patients continue to receive ADT and receive testosterone cypionate intramuscularly (IM) on day 1 of cycles 1-6. Patients receive LuPSMA IV on day 1 of cycles 2-6. Cycles repeat every 6 weeks for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive testosterone cypionate intramuscularly (IM) on day 1 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo 68Ga-PSMA positron emission tomography (PET) at screening and single photon emission computed tomography (SPECT)/CT throughout the study.

COHORT IIIb: Patients continue to receive ADT and LuPSMA IV on day 1 of cycles 1-6. Patients also receive receive testosterone cypionate IM on day 1 of cycles 2-6 . Cycles repeat every 6 weeks for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients receive testosterone cypionate IM on day 1 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo 68Ga-PSMA PET at screening and single SPECT/CT throughout the study.

COHORT IIIc: Patients continue to receive ADT and receive testosterone cypionate IM on day 1 and LuPSMA IV on day 1 of cycles 1-6. Cycles repeat every 6 weeks for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive testosterone cypionate IM on day 1 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo 68Ga-PSMA PET at screening and single SPECT/CT throughout the study.

All patients undergo a biopsy on study and blood sample collection on study, and bone scans, dual x-ray absorptiometry (DEXA) and computed tomography (CT) scans throughout the trial. Patients may also undergo an optional second biopsy at the end of study treatment.

After completion of study treatment, patients are followed up at 30 days, and then every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Must be willing to provide informed consent prior to any study specific procedures
* Age >= 18 years
* Documented histologically confirmed adenocarcinoma of the prostate
* Patient must have evidence of castration resistant prostate cancer as evidenced by PSA progression (per Prostate Cancer Working Group 3 [PCWG3] criteria) and a castrate serum testosterone level (i.e., =< 50 mg/dL)
* PSA must be at least 2 ng/ml and rising on two successive measurements at least two weeks apart
* Patients must have progressed on at least one prior next-generation androgen receptor-signalling inhibitor (e.g., abiraterone, enzalutamide, etc.). There must be at least a 2-week washout period after stopping the most recent approved therapy for metastatic castration-resistant prostate cancer (mCRPC) (e.g., abiraterone, enzalutamide, Ra-223, sipuleucel-t) prior to cycle 1, day 1. If applicable, patients should be weaned off steroids at least 1 week prior to starting treatment
* Subjects enrolling to Cohort 3 must demonstrate evidence of PSMA expression on 68Ga-PSMA-11 PET as defined in the VISION trial
* No prior chemotherapy for the treatment of mCRPC. Patients may have received docetaxel for the treatment of hormone-sensitive prostate cancer
* Prior treatment with non-chemotherapy investigational agents is permitted. There must be at least a 2-week washout period after stopping any investigational cancer agent prior to cycle 1, day 1
* Hemoglobin >= 9 g/dL with no blood transfusion in the past 28 days (within 30 days prior to administration of study treatment)
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L (within 30 days prior to administration of study treatment)
* Platelet count >= 100 x 10^9/L (within 30 days prior to administration of study treatment)
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (within 30 days prior to administration of study treatment)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) / alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal unless liver metastases are present in which case they must be =< 5x ULN (within 30 days prior to administration of study treatment)
* Patients must have creatinine clearance estimated using the Cockcroft-Gault equation or based on 24 hour urine test of >= 51 mL/min (within 30 days prior to administration of study treatment)
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Patients must have a life expectancy >= 16 weeks
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations
* At least one lesion (measurable and/or non-measurable) that can be accurately assessed at baseline by CT, positron emission tomography (PET), magnetic resonance imaging (MRI) and/or bone scan and is suitable for repeated assessment
* Must be willing to undergo metastatic biopsy and have a lesion amenable for biopsy
* Male patients and their partners, who are sexually active and of childbearing potential, must agree to the use of two highly effective forms of contraception in combination, throughout the period of taking study treatment and for 6 months after last dose of study drug(s) to prevent pregnancy in a partner

Exclusion Criteria:

* Involvement in the planning and/or conduct of the study
* Other malignancy unless curatively treated with no evidence of disease for >= 2 years except: adequately treated non-melanoma skin cancer, non-muscle invasive bladder cancer
* Persistent toxicities (Common Terminology Criteria for Adverse Event (CTCAE) grade > 2) caused by previous cancer therapy, excluding alopecia
* Patients with symptomatic uncontrolled brain metastases. A scan to confirm the absence of brain metastases is not required. Patients with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease for 28 days
* Use of corticosteroids at a dose equivalent to > 10 mg of prednisone daily
* Planning to receive concurrent treatment with another systemic cancer therapy, aside from a luteinizing hormone releasing hormone (LHRH) analogue
* Use of warfarin is not permitted. Low-molecular weight heparin and direct oral anticoagulants are allowed, but their use should be discussed with the principal investigator (PI) first
* Major surgery within 2 weeks of starting study treatment and patients must have recovered from any effects of any major surgery
* Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, uncontrolled major seizure disorder, uncontrolled hypertension (blood pressure [BP] >= 165/100), history of prior stroke, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease or any psychiatric disorder that prohibits obtaining informed consent
* Patients with a known hypersensitivity to the testosterone cypionate, etoposide, carboplatin or any of the excipients of these products
* Patients with known active hepatitis (i.e., hepatitis B or C) due to risk of transmitting the infection through blood or other body fluids
* Evidence of serious and/or unstable pre-existing medical, psychiatric or other condition (including laboratory abnormalities) that could interfere with patient safety or provision of informed consent to participate in this study
* Any psychological, familial, sociological, or geographical condition that could potentially interfere with compliance with the study protocol and follow-up schedule
* Evidence of disease that, in the opinion of the investigator, would put the patient at risk from testosterone therapy (e.g. femoral metastases with concern over fracture risk, spinal metastases with concern over spinal cord compression, lymph node disease with concern for ureteral obstruction)
* Patients with pain attributable to their prostate cancer.

  * Excluded due to concern for pain flare due to testosterone supplementation
* Tumor causing urinary outlet obstruction that requires catheterization for voiding. Patients that require catheterization to void secondary to benign strictures or other non-cancer causes will be permitted to enroll. Patients with percutaneous nephrostomy tubes will also be permitted to enroll
* Prior history of deep venous thrombosis or pulmonary embolism within 5 years prior to enrollment in the study and not currently on systemic anticoagulation.

  * Excluded due to risk of venous thromboembolism from hormone supplementation
* Patients with NYHA (New York Heart Association) class III or IV heart failure or history of a prior myocardial infarction (MI) within 5 years of enrollment to the study.

  * Excluded due to increased risk of cardiovascular events with testosterone supplementation

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2024-05-21 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Greater than or equal to 50% decline in prostate-specific antigen from baseline (PSA50) response rate | From baseline up to 3 years
  Will assess >= 50% decline in PSA following treatment with combination bipolar androgen therapy (BAT) and genotoxic chemotherapy (at least 12 weeks of total therapy). Will be calculated as the percentage with 95% confidence interval (CI) of the total number of subjects that achieved a PSA50 response.

SECONDARY OUTCOMES:
Radiographic response | Up to 3 years
  Will be assessed using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Best radiographic response for each patient will be presented in a waterfall plot.
Radiographic progression-free survival (PFS) | The start of treatment until disease progression (per modified RECIST criteria or PCWG3 criteria for bone lesions), clinical progression (as determined by the treating physician), or death, whichever occurs first, assessed up to 3 years
  Will be assessed using RECIST 1.1 and Prostate Cancer Working Group 3 (PCWG3) criteria. Will be presented with Kaplan-Meier curves, and the median survival with 95% CI will be calculated. Rates will be reported as percentages with 95% CI.
PSA PFS | Time from the start of treatment until PSA progression (as defined by PCWG3 criteria), assessed up to 3 years
  Will be assessed using PCWG3 criteria. Will be presented with Kaplan-Meier curves, and the median survival with 95% CI will be calculated. Rates will be reported as percentages with 95% CI. Best on study PSA for each patient will be presented in a waterfall plot.
Overall survival | The start of treatment until death from any cause, assessed up to 3 years
  Will be presented with Kaplan-Meier curves, and the median survival with 95% CI will be calculated. Rates will be reported as percentages with 95% CI.
Patient-reported outcome measure (PROMS) questionnaires | Up to 3 years
  Will be assessed by average change in quality of life (QOL) scores (total and for each domain) for each survey will be calculated at each timepoint. A paired t-test will used to assess for statistically significant changes in QOL from baseline to subsequent timepoints, and linear mixed effects models will be used to evaluate trends over all timepoints.
Incidence of adverse events | Up to 30 days after completion of study treatment
  Will be assessed according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Schweizer, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No